CLINICAL TRIAL: NCT04481061
Title: Engaging Adolescents in Decisions About Return of Genomic Research Results
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5R01HG010166-02 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Genetic Screening; Adolescent; Genetic Change; Shared Decision Making; Knowledge, Attitudes, Practice; Genetic Testing
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Adolescents between 13-21 years of age will be given the option to learn categories of genomic results. Results will be returned based on their choices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Making About Genetic Results (Other): Adolescents between 13-21 and parent (if applicable) will make decisions about learning results using an electronic decision tool. Results that match their choices will be returned.
  Interventions: Genetic: Electronic Decision Tool

INTERVENTIONS:
Genetic: Electronic Decision Tool — Adolescents and a parent, if applicable, will use an electronic decision tool to make categorical choices of types of diseases (treatable, preventable, adult-onset, and carrier status) they want to learn about the adolescent. Granular choices can be made within each category.

SUMMARY:
Recent recommendations to return children's results for adult-onset conditions to parents anytime whole exome or genome sequencing is performed, as well as growing expectations to return research results to participants on a large-scale basis, mean adolescents will increasingly be engaged in assenting (<age 18) and consenting (>age 18) to return of genomic research results. There is an urgent need to understand adolescents' informational preferences and to create ethically informed, scalable processes that empower adolescents from diverse backgrounds to participate in the decision-making process about learning genomic results. This research will provide important insights into adolescents' choices, as well as the ethical, legal and societal implications of engaging adolescents in making choices about learning genomic results in genomic research and community-based research settings.

DETAILED DESCRIPTION:
The purpose of this study is to assess assenting and consenting adolescents' choices about learning genomic research results. The investigator will refine existing decision tools and processes to promote informed genomic decision-making through the use of focus groups with adolescents and parents recruited from an existing genomic research study and a diverse, medically-underserved community to assess whether and how recruitment pathways impact perceived value, risks, and benefits of participation in genomic research and return of personal genomic information. Once these materials have been refined, consenting adolescents between the ages of 18-21, assenting adolescents between the ages of 13-17, and their parents (optional for consenting adolescents) will be invited to make choices using an electronic decision tool for an actual return of results study using two different genome sequencing panels. A joint decision-making process involving adolescents, a parent (if applicable), and a study team member will facilitate confirmation of choices. A subset of adolescents will also be asked to reflect upon the genetic results they chose to learn, factors that impacted their choices, and decision-stability during in-depth interviews. Genomic research results will be returned that reflect the participants' choices. Surveys and interviews will be conducted following return of results to assess participants' understanding, perceived risks and benefits, psychosocial and behavioral impact, and whether decisional regret is associated with decisional stability. Throughout the study legal, ethical, and social issues pertaining to adolescents' preferences and responses to return of genomic research results will be explored, including normative assessments of empirical findings as well as the population-level utility and impact of involving adolescents in the decision-making process. Findings from this study will contribute to filling a critical gap in the literature regarding engaging adolescents' in the decision to learn genomic research results, and will help inform best practices with adolescent populations. This information is critical given recent recommendations by the American College of Medical Genetics to return children's results for adult onset conditions to parents' anytime whole exome or genome sequencing is performed. Findings from this study will also help inform a growing expectation to return research results on a large-scale basis, necessitating examination of ethical return of research results with a range of populations recruited from a variety of settings.

ELIGIBILITY:
Inclusion Criteria:

* Assenting adolescents (13-17 years)
* Consenting adolescents (18-21 years)
* Parent / legal guardian of assenting or consenting adolescent
* Ability to participate in remote study visits, if applicable

Exclusion Criteria:

* Those who do not meet inclusion criteria
* Those who do not communicate in English
* Individuals with developmental disabilities that interfere with their ability to make independent decisions

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Participant Choices Throughout the Study | Pre-intervention baseline choices made at enrollment; choices made during the intervention (about one hour after baseline); post-intervention choices (4 weeks after intervention); post return of results choices (an average of 1 year after intervention).
  Choices will be operationalized as the decisions to receive all results, some results, or no results. We will be measuring the changes in these choices at various time points, including from baseline to immediately after the intervention (about one hour after baseline), and again four weeks after the intervention.
Change in Participant's "Decisional Conflict Scale" Score Throughout the Study | Decisional Conflict will be measured at baseline, immediately after the intervention (about one hour after baseline), and four weeks after the intervention.
  Decisional conflict is a continuous variable measured using a validated scale called the Decisional Conflict Scale. Decisional conflict will vary depending on the difficulty of the decision being made and is greater if an individual feels uninformed about benefits and risks of a decision, is unclear about their values, or feels unsupported or pressured to make a decision. The scale will range from 0-100. The more conflicted someone is the higher the score.
Change in Participant Decisional Stability Throughout the Study | Measured at baseline, immediately after the intervention, (within an hour of baseline), and four weeks after the intervention.
  Decisional stability will be measured by the proportion of assenting and consenting adolescents whose choices stay consistent or change at the three time points (baseline, immediately after the intervention, four weeks after the intervention)
Measurement of Participant's Post Return of Results Decision Regret Score | Measurement taken within one week after returning results. This is an average of 1 year of the intervention.
  The "Decision Regret Scale" is a validated scale that measures distress or remorse after a healthcare decision. The scale ranges from 0- 100. The higher the score, the more the person regrets their choices.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Michelle McGowan, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Blumling AA, McGowan ML, Prows CA, Childers-Buschle K, Martin LJ, Lynch JA, Dufendach KR, Lipstein EA, Kovacic MB, Brinkman WB, Myers MF. Engaging adolescents and young adults in decisions about return of genomic research results: study protocol for a mixed-methods longitudinal clinical trial protocol. BMC Med Inform Decis Mak. 2024 Dec 18;24(1):391. doi: 10.1186/s12911-024-02784-w. PMID 39696322

DOCUMENTS (3):
  • Informed Consent Form: Parental Permission_Adult Consent (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04481061/ICF_000.pdf
  • Informed Consent Form: Consent Young Adult (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04481061/ICF_001.pdf
  • Informed Consent Form: Assent (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04481061/ICF_002.pdf